CLINICAL TRIAL: NCT00001379
Title: Treatment and Natural History Study of Lymphomatoid Granulomatosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christopher Melani, MD, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 940074; 94-C-0074; NCT00018993 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Lymphomatoid Granulomatosis; Granulomatosis, Lymphomatoid; Non-Hodgkins Lymphoma; Lymphoproliferative Disorder
Keywords: Epstein-Barr Virus; Lymphoproliferative Disorder; Viral; Immunosuppression; Lymphoma
MeSH Terms: conditions — Lymphomatoid Granulomatosis; Lymphoma, Non-Hodgkin; Lymphoproliferative Disorders; Epstein-Barr Virus Infections; Lymphoma | interventions — Interferons; Rituximab; EPOCH protocol; Etoposide; Prednisone; Vincristine; Cyclophosphamide; Doxorubicin; Tomography, X-Ray Computed; Echocardiography; Caves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1-Interferon (Experimental): Interferon starting at 7.5 million Units subcutaneous (subQ) 3 times a week and increasing on the designated schedule, as tolerated. Patients continue taking interferon for 1 year beyond complete remission (CR). Patients who progress may crossover to receive etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin and rituximab (EPOCH-R).
  Interventions: Biological: Interferon; Procedure: Tumor biopsy; Procedure: Bone marrow biopsy; Biological: Bone marrow aspirate; Procedure: Lumber puncture; Diagnostic Test: CT; Diagnostic Test: Brain MRI; Diagnostic Test: Echocardiogram; Diagnostic Test: FDG-PET
- Arm 2-Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab (EPOCH-R) (Experimental): Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin and rituximab (EPOCH-R) every 3 weeks for up to 6 cycles, based on response. Participants who relapse or progress may crossover to receive interferon.
  Interventions: Drug: Rituxan and EPOCH; Procedure: Tumor biopsy; Procedure: Bone marrow biopsy; Biological: Bone marrow aspirate; Procedure: Lumber puncture; Diagnostic Test: CT; Diagnostic Test: Brain MRI; Diagnostic Test: Echocardiogram; Diagnostic Test: FDG-PET

INTERVENTIONS:
Biological: Interferon — For lymphomatoid granulomatosis (LYG) Grade 1 and 2: Interferon starting at 7.5 million Units subcutaneous (subQ) 3 times a week and increasing on the following schedule: 10 million U; 15 million U; 20 million U; 25 million U; and increased in 5 million U increments, as tolerated. Patients continue taking interferon for 1 year beyond complete remission (CR).
  Other Names: IFN
  Arms: Arm 1-Interferon
Drug: Rituxan and EPOCH — For lymphomatoid granulomatosis (LYG) Grade 3: EPOCH-R (etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, rituximab) every 3 weeks for 6 cycles.
  Other Names: Rituximab; etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, rituximab
  Arms: Arm 2-Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin & Rituximab (EPOCH-R)
Procedure: Tumor biopsy — Baseline (optional).
  Other Names: Tumor bx
Procedure: Bone marrow biopsy — Baseline.
  Other Names: BM biopsy
Biological: Bone marrow aspirate — Baseline.
  Other Names: BM aspirate
Procedure: Lumber puncture — Baseline.
  Other Names: LP
Diagnostic Test: CT — Arm 1: At baseline, then every 4 weeks until on stable dose of interferon or a maximum of 6 monthly scans, then every 3 months while receiving interferon, and following completion of interferon. In surveillance, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year and yearly thereafter for 2 years. Arm 2: At baseline, following cycle 4, and following cycle 6 of etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (DA-EPOCH-R). In surveillance, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year and yearly thereafter for 2 years.
  Other Names: Computed tomography
Diagnostic Test: Brain MRI — Arm 1: At baseline, then every 4 weeks until on stable dose of interferon or a maximum of 6 monthly scans, then every 3 months while receiving interferon, and following completion of interferon. In surveillance, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year and yearly thereafter for 2 years (patients with central nervous system (CNS) disease only).
  Arm 2: At baseline, following cycle 4, and following cycle 6 of etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (DA-EPOCH-R). In surveillance, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year and yearly thereafter for 2 years (patients with CNS disease only).
  Other Names: Brain magnetic resonance imaging
Diagnostic Test: Echocardiogram — For participants receiving > 450 mg/m^2 doxorubicin.
  Other Names: Echo
Diagnostic Test: FDG-PET — Arm 1: Baseline and following completion of interferon. Arm 2: Baseline and following completion of etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (DA-EPOCH-R).
  Other Names: Fluorodeoxyglucose positron emission tomography

SUMMARY:
This study will evaluate the response and long-term effects of alpha-interferon in patients with lymphomatoid granulomatosis (LYG). The disease causes proliferation of destructive cells involving the lungs, skin, kidneys, and central nervous system.

Patients ages 12 and older who have LYG and who are not pregnant, or breast feeding may be eligible for this study. Alpha interferon or chemotherapy, or both, will be used. Alpha interferon is a protein the body naturally produces. If patients have grade 3 disease, they will usually receive etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin (EPOCH)-rituximab (EPOCH-R) chemotherapy (each letter representing a drug). If patients have grade 1 or 2 disease, they will usually receive alpha interferon. If patients have LYG after receiving alpha interferon and/or EPOCH-R, they may receive rituximab alone or with alpha interferon. Rituximab is an antibody, binding to a specific molecule cluster of differentiation 20 (CD20) present on most B-cell lymphomas. Doses of several drugs in EPOCH-R may be increased if patients tolerated them in the previous cycle. If patients respond to EPOCH-R but still have low grade LYG, they may receive alpha interferon. Researchers will also try to obtain a biopsy of patient's lesions, to help in understanding the disease.

Patients self-administer alpha interferon by injection under the skin three times weekly. They will visit the clinic every 2 to 12 weeks for follow-up. Patients will receive alpha interferon for 1 year after LYG goes away, depending on response. EPOCH-R has these drugs: rituximab by vein on Day 1; prednisone by mouth on Days 1 to 5; etoposide, doxorubicin, and vincristine as a continuous intravenous infusion on Days 1 to 5; and cyclophosphamide by intravenous injection over 1 hour on Day 5. Each cycle lasts 3 weeks: 5 days of chemotherapy and 16 days of no chemotherapy. Etoposide, doxorubicin, and vincristine are infused through a small pump worn by patients. The drugs are given over 5 days through a central intravenous catheter. There are two cycles of EPOCH-R beyond a maximum response, with six cycles maximum. To reduce harm to bone marrow, patients receive granulocyte colony stimulating factor (G-CSF), self-administered by injection under the skin daily for approximately 10 days between chemotherapy cycles. If at the end of therapy, patients have a complete response, treatment will stop. If there is residual low-grade disease, patients may receive alpha interferon. Alpha interferon can have flu-like side effects of headache, fever, chills, and body aches. EPOCH-R drugs can cause gastrointestinal problems, hair loss, and weakness. Granulocyte colony-stimulating factor (G-CSF) can cause bone pain, body aches, and hair thinning. Chemotherapy can cause some patients to develop leukemia.

This study may or may not have a direct benefit for participants. It is not certain whether the new therapy will help decrease tumors. However, knowledge gained may improve the understanding of and treatment for LYG.

...

DETAILED DESCRIPTION:
BACKGROUND:

* Lymphomatoid granulomatosis (LYG) is an angiocentric destructive proliferation of lymphoid cells predominantly involving the lungs, skin, kidneys, and central nervous system.
* It is divided into three grades, depending on the degree of necrosis and cellular atypia. The grades of disease are histologically based and do not necessarily correlate with clinical outcome. However, like other Epstein-Barr virus (EBV) related lymphoproliferative disorders (LPD's), LYG can transform into an aggressive large B-cell lymphoma, which would be included within the grade 3 category. It is important to note that not all grade 3 lesions are a large B-cell lymphoma.
* Current evidence shows that LYG is a disease of B cells.

OBJECTIVES:

* To determine the response and long-term efficacy of alpha-Interferon in patients with lymphomatoid granulomatosis (LYG).
* To determine the response and long-term efficacy of dose-adjusted (DA)-etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin rituximab (EPOCH-R) chemotherapy in patients with grade 3 LYG or in patients who have failed interferon.

ELIGIBILITY:

* Patients must have a tissue diagnosis of grade 1, 2 and/or 3 LYG (or a diagnosis consistent with LYG) confirmed by the Laboratory of Pathology, National Cancer Institute (NCI).
* Patients with any stage of disease will be eligible.
* Previously untreated and treated patients are eligible.
* Patients aged 12 or older will be eligible.

DESIGN:

* Interferon is used as initial treatment in patients with grades 1 and 2 LYG. Patients will receive interferon for one year past complete remission (CR).
* Patients who progress after or during interferon, and patients with grade 3 LYG will receive aggressive combination chemotherapy with DA-EPOCH-R (rituximab, etoposide, doxorubicin, vincristine, cyclophosphamide and prednisone).
* Patients who fail one treatment approach may be crossed over to the other.
* A total of 105 patients will be enrolled at this single institution.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have a tissue-diagnosis of grade 1, 2 and/or 3 lymphomatoid granulomatosis (LYG) (or a diagnosis consistent with LYG) confirmed by the Laboratory of Pathology, National Cancer Institute (NCI). Final histopathologic classification and pathologic grade will be determined by Stephania Pittaluga, medical doctor (M.D.) or her designee.

Patients with any stage of disease will be eligible.

Previously untreated and treated patients are eligible.

Patients aged 12 or older will be eligible.

EXCLUSION CRITERIA:

Patients with a history of coronary artery disease with angina pectoris, or a history of congestive heart failure will not be eligible to receive. etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin and rituximab (DA-EPOCH-R) chemotherapy.

Patients with significant renal (serum creatinine (Cr.) greater than 1.5 mg/dl or creatinine clearance less than 40 cc/min) or hepatic (bilirubin greater than 2.5 x upper limit of normal (ULN) dysfunction not due to tumor involvement will not be eligible to receive DA-EPOCH-R chemotherapy.

Informed consent must be obtained.

Patients who in the opinion of the principal investigator are poor psychiatric or medical risk are not eligible.

Patients who received > 450 mg/m^2 doxorubicin and have a cardiac ejection fraction on echocardiogram less than or equal to 40% on protocol entry are not eligible to received DA-EPOCH-R.

Patients with prior hepatitis B exposure may be included in the study provided that they have hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels below the World Health Organizations cutoff of 100 IU/mL prior to starting therapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 1995-05-05 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Melani, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Derived] Melani C, Dowdell K, Pittaluga S, Dunleavy K, Roschewski M, Song JY, Calattini S, Kawada JI, Price DA, Chattopadhyay PK, Roederer M, Lucas AN, Steinberg SM, Jaffe ES, Cohen JI, Wilson WH. Interferon alfa-2b in patients with low-grade lymphomatoid granulomatosis and chemotherapy with DA-EPOCH-R in patients with high-grade lymphomatoid granulomatosis: an open-label, single-centre, phase 2 trial. Lancet Haematol. 2023 May;10(5):e346-e358. doi: 10.1016/S2352-3026(23)00029-7. Epub 2023 Mar 31. PMID 37011643
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1994-C-0074.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Treated With Initial Interferon Therapy: Interferon starting at 7.5 million Units subcutaneous (subQ) 3 times a week and increasing on the designated schedule, as tolerated. Participants continue taking interferon for 1 year beyond complete remission (CR). Patients who progress may crossover to receive etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin and rituximab (EPOCH-R).
  Interferon: For lymphomatoid granulomatosis (LYG) Grade 1 and 2: Interferon starting at 7.5 million Units subcutaneous (subQ) 3 times a week and increasing on the following schedule: 10 million U; 15 million U; 20 million U; 25 million U; and increased in 5 million U increments, as tolerated. Participants continue taking interferon for 1 year beyond complete remission (CR).
- Treated With Initial Etoposide,Prednisone,Vincristine,Cyclophosphamide,Doxorubicin,Rituximab Therapy: Etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin and rituximab (EPOCH-R) every 3 weeks for up to 6 cycles, based on response.
  Rituxan and EPOCH: For lymphomatoid granulomatosis (LYG) Grade 3: EPOCH-R (etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, rituximab) every 3 weeks for 6 cycles.
  Participants who relapse or progress may crossover to receive interferon.
- Participants Enrolled But Not Treated: Participants were enrolled and not treated with initial interferon or etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin and rituximab (EPOCH-R) therapy.
- Participant Treated With Rituximab and Radiation Only: Participant treated with rituximab and radiation only. Did not receive either interferon or etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R) therapy.
Period: Initial Treatment
Arm/Group | Participants Treated With Initial Interferon Therapy | Treated With Initial Etoposide,Prednisone,Vincristine,Cyclophosphamide,Doxorubicin,Rituximab Therapy | Participants Enrolled But Not Treated | Participant Treated With Rituximab and Radiation Only
Started | 60 | 28 | 5 | 1
Participants Eligible for Cross-over to EPOCH-R | 24 | 0 | 0 | 0
Participants Eligible for Cross-over to Interferon | 0 | 10 | 0 | 0
Participants Did Not Cross Over to Interferon or EPOCH Therapy After Initial Treatment | 36 | 18 | 0 (Did not receive initial therapy with interferon or EPOCH-R.) | 0 (Did not receive initial therapy with interferon or EPOCH-R.)
Completed | 29 | 23 | 0 | 0
Not Completed | 31 | 5 | 5 | 1
Not completed — Disease progression | 21 | 3 | 0 | 0
Not completed — Complicating disease/intercurrent illness | 6 | 1 | 0 | 0
Not completed — Received alternative treatment | 2 | 1 | 0 | 0
Not completed — Refused further treatment | 2 | 0 | 0 | 0
Not completed — Did not receive protocol treatment | 0 | 0 | 5 | 0
Not completed — Received treatment with whole brain radiation therapy (WBRT) + Rituximab | 0 | 0 | 0 | 1
Period: Cross-Over After Initial Treatment
Arm/Group | Participants Treated With Initial Interferon Therapy | Treated With Initial Etoposide,Prednisone,Vincristine,Cyclophosphamide,Doxorubicin,Rituximab Therapy | Participants Enrolled But Not Treated | Participant Treated With Rituximab and Radiation Only
Started | 24 | 10 | 0 | 0
Participants Eligible for Cross-over Treated With EPOCH-R | 24 | 0 | 0 | 0
Participants Eligible for Cross-over Treated With Interferon | 0 | 10 | 0 | 0
Completed | 14 | 7 | 0 | 0
Not Completed | 10 | 3 | 0 | 0
Not completed — Disease progression | 4 | 2 | 0 | 0
Not completed — Complicating disease/intercurrent illness | 1 | 1 | 0 | 0
Not completed — Received alternative treatment | 4 | 0 | 0 | 0
Not completed — Refused further treatment | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data collected for 5 participants who were enrolled and not treated are reported here.
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Treated With Initial Interferon Therapy | Treated With Initial Etoposide,Prednisone,Vincristine,Cyclophosphamide,Doxorubicin,Rituximab Therapy | Participants Enrolled But Not Treated | Participant Treated With Rituximab and Radiation Only | Total
Number analyzed (Participants) | 60 | 28 | 5 | 1 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 0 | 0 | 2
  Between 18 and 65 years | 54 | 27 | 5 | 1 | 87
  >=65 years | 5 | 0 | 0 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (13.88) | 47.42 (12.76) | 42.64 (12.47) | 18 (0) | 46.33 (13.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 14 | 2 | 1 | 38
  Male | 39 | 14 | 3 | 0 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 60 | 28 | 5 | 1 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 3 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 0 | 2
  White | 53 | 25 | 5 | 1 | 84
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 0 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 60 | 28 | 5 | 1 | 94
Baseline Histologic Grade of Lymphomatoid Granulomatosis (LYG) [Count of Participants; unit: Participants] — Grade 1 LYG is rare atypical lymphoid cells, Epstein Barr virus-encoded ribonucleic acid (EBER)(+) cells, typically <5 cells/high-power field (HPF), and focal to absent necrosis. Grade 2 LYG has a greater number of large atypical lymphoid cells, EBER+ cells between 5-20 and occasionally up to 50 cells/HPF, and often extensive necrosis. Grade 3 LYG has a greater number of large atypical lymphoid cells, EBER+ cells typically >50 and often >100 cells/HPF, and often extensive necrosis. Not applicable (NA) = These were not graded due to having an alternative diagnosis other than LYG.
  Participants
    Grade 1 | 22 | 1 | 0 | 0 | 23
    Grade 2 | 19 | 2 | 1 | 0 | 22
    Grade 3 | 13 | 22 | 2 | 0 | 37
    NA | 6 | 3 | 2 | 1 | 12
Prior Therapy [Count of Participants; unit: Participants] — Categories of therapy are not mutually exclusive.
  Participants
    None | 16 | 13 | 1 | 0 | 30
    Corticosteroids | 42 | 14 | 3 | 1 | 60
    Chemotherapy | 22 | 4 | 2 | 1 | 29
    Rituximab | 13 | 3 | 3 | 0 | 19
Disease Sites [Count of Participants; unit: Participants] — Other = sinus/nasal cavity, prostate, eyelid/conjunctiva, muscle, pancreas, vertebrae, vocal cord, parotid gland, and stomach). Categories are not mutually exclusive.
  Participants
    Lung | 60 | 28 | 5 | 0 | 93
    Central nervous system (CNS) | 21 | 8 | 0 | 1 | 30
    Skin | 20 | 11 | 1 | 0 | 32
    Kidney | 11 | 4 | 0 | 0 | 15
    Liver | 10 | 6 | 1 | 0 | 17
    Spleen | 6 | 3 | 1 | 0 | 10
    Lymph node | 4 | 1 | 0 | 0 | 5
    Other | 9 | 9 | 2 | 0 | 20
Elevated lactate hydrogenase (LDH) [Count of Participants; unit: Participants] | 31 | 12 | 2 | 0 | 45
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Performance status 0 is normal activity, fully active, able to carry on all pre-disease performance without restriction. 1 is symptoms but ambulatory, restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. 2 is in bed <50% of the time, ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours. 3 is in bed >50% of the time, capable of only limited self-care, confined to bed or chair more than 50% of waking hours. 4 is 100% bedridden. Performance status 5 is dead.
  Participants
    0-1 | 47 | 24 | 5 | 1 | 77
    ≥2 | 13 | 4 | 0 | 0 | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate will be classified as the following: complete remission (CR), partial remission (PR), disease progression or disease stabilization measured by the Response Criteria. CR is no evidence of active disease on restaging for at least 2 months duration. All lesions must have decreased by > 75%, be gallium or positron emission tomography (PET) negative (if obtained) and be stable for > 3 months without new lesions appearing. PR is 50% or greater decrease in the sum of the products of the diameters of all measurable lesions for at least one month. Disease progression is 25% or greater progression in the sum of the products of the diameter of any measurable lesion over one month or the appearance or any new lesion consistent with metastatic disease. Disease stabilization is no change in the sum of the products of the diameters of all measurable lesions over two months and no new lesions consistent with disease.
Time Frame: From study enrollment and throughout treatment, up to a maximum of 40 months for the 2 interferon groups and 8 months for the 2 EPOCH-R groups.
Population: 9/94 participants were not analyzed because 5 were enrolled and not treated,3 participants died prior to restaging scans, and 1 was treated with rituximab and radiation only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treated With Interferon&Crossed Over - Prednisone,Vincristine,Cyclophosphamide,Doxorubicin,Rituximab: All participants who were treated with initial interferon and crossed over to receive etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R).
- Treated With Pednisone,Vincristine,Cyclophosphamide,Doxorubicin,Rituximab&Crossed Over to Interferon: All participants who were treated with initial prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R) and crossed over to receive interferon.
Arm/Group | Participants Treated With Initial Interferon Therapy | Treated With Initial Etoposide,Prednisone,Vincristine,Cyclophosphamide,Doxorubicin,Rituximab Therapy | Treated With Interferon&Crossed Over - Prednisone,Vincristine,Cyclophosphamide,Doxorubicin,Rituximab | Treated With Pednisone,Vincristine,Cyclophosphamide,Doxorubicin,Rituximab&Crossed Over to Interferon
Number analyzed (Participants) | 58 | 27 | 21 | 10
percentage of participants
  Complete Remission | 53.45 [40.80 to 65.67] | 51.85 [33.99 to 69.26] | 57.14 [36.55 to 75.53] | 50.00 [23.66 to 76.34]
  Partial Remission | 5.17 [1.14 to 14.14] | 25.93 [13.17 to 44.68] | 14.29 [4.98 to 34.64] | 10.00 [0.51 to 40.12]
  Disease Progression | 32.76 [22.08 to 45.58] | 11.11 [3.85 to 28.06] | 14.29 [4.98 to 34.64] | 20.00 [3.55 to 50.98]
  Disease Stabilization | 8.62 [3.74 to 18.64] | 11.11 [3.85 to 28.06] | 14.29 [4.98 to 34.64] | 20.00 [3.55 to 50.98]

2. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from the date of study enrollment until the date of disease relapse, disease progression, death, or last follow-up, whichever occurs first, using the Kaplan-Meier method. Response was assessed by the Lugano Classification Response Criteria for Non-Hodgkin lymphoma (NHL). Disease progression is defined as an increase of ≥ 50% from the product of the perpendicular diameter (PPD) nadir and an increase in longest transverse diameter of a lesion (LDi) or shortest axis perpendicular diameter (SDi) from nadir of >0.5 cm for lesions <2 cm or >1.0 cm for lesions >2 cm.
Time Frame: Assessed from date of study enrollment until time of disease relapse, disease progression, death, or last follow-up, whichever comes first, up to a maximum of 27 years for the 2 interferon groups and 20 years for the 2 EPOCH-R groups.
Population: 6/94 participants were not analyzed because 5 were enrolled and not treated, and 1 was treated with rituximab and radiation only.
Measure: Median (95% Confidence Interval); unit: years
Groups:
- Treated With Initial Interferon Therapy: Interferon starting at 7.5 million Units subcutaneous (subQ) 3 times a week and increasing on the designated schedule, as tolerated. Participants continue taking interferon for 1 year beyond complete remission (CR). Patients who progress may crossover to receive etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin and rituximab (EPOCH-R).
  Interferon: For lymphomatoid granulomatosis (LYG) Grade 1 and 2: Interferon starting at 7.5 million Units subcutaneous (subQ) 3 times a week and increasing on the following schedule: 10 million U; 15 million U; 20 million U; 25 million U; and increased in 5 million U increments, as tolerated. Participants continue taking interferon for 1 year beyond complete remission (CR).
Arm/Group | Treated With Initial Interferon Therapy | Treated With Initial Etoposide,Prednisone,Vincristine,Cyclophosphamide,Doxorubicin,Rituximab Therapy | Treated With Interferon&Crossed Over - Prednisone,Vincristine,Cyclophosphamide,Doxorubicin,Rituximab | Treated With Pednisone,Vincristine,Cyclophosphamide,Doxorubicin,Rituximab&Crossed Over to Interferon
Number analyzed (Participants) | 60 | 28 | 24 | 10
years | 1.01 [0.61 to 6.54] | 0.69 [0.45 to 8.43] | 0.23 [0.14 to 0.49] | 0.53 [0.33 to NA] — Confidence intervals are generated via the Brookmeyer-Crowley method (if a limit of the confidence interval does not intersect the median, then it is recorded as not estimable (i.e., NA).

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from treatment start date until date of death or date last known alive. The median OS will be determined and reported along with a 95% confidence interval.
Time Frame: Assessed from date of study enrollment until time of death or last follow-up, whichever comes first, up to a maximum of 27 years.
Population: 6/94 participants were not analyzed because 5 were enrolled and not treated and 1 was treated with rituximab and radiation only.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Participants Treated With Initial Interferon Therapy | Treated With Initial Etoposide,Prednisone,Vincristine,Cyclophosphamide,Doxorubicin,Rituximab Therapy | Treated With Interferon&Crossed Over - Prednisone,Vincristine,Cyclophosphamide,Doxorubicin,Rituximab | Treated With Pednisone,Vincristine,Cyclophosphamide,Doxorubicin,Rituximab&Crossed Over to Interferon
Number analyzed (Participants) | 60 | 28 | 24 | 10
years | 12.22 [7.29 to NA] — Confidence intervals are generated via the Brookmeyer-Crowley method (if a limit of the confidence interval does not intersect the median, then it is recorded as not estimable (i.e., NA). | 9.84 [3.35 to NA] — Confidence intervals are generated via the Brookmeyer-Crowley method (if a limit of the confidence interval does not intersect the median, then it is recorded as not estimable (i.e., NA). | 8.43 [2.66 to NA] — Confidence intervals are generated via the Brookmeyer-Crowley method (if a limit of the confidence interval does not intersect the median, then it is recorded as not estimable (i.e., NA). | 12.13 [2.89 to NA] — Confidence intervals are generated via the Brookmeyer-Crowley method (if a limit of the confidence interval does not intersect the median, then it is recorded as not estimable (i.e., NA).

4. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Toxicity Criteria (CTC v2.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Toxicity Criteria (CTC v2.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Adverse Events were monitored/assessed from the first study intervention, Study Day 1 of Cycle 1 through 30 days after the study agent (s) was/were administered, up to a maximum of 49 months.
Population: 5 participants who were followed and not treated on study were followed for survival and mortality.
Measure: Count of Participants; unit: Participants
Groups:
- Participants Enrolled But Not Treated: Participants were enrolled and not treated with initial interferon or etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin and rituximab (EPOCH-R) therapy.
  5 participants were followed and not treated on study were followed for survival and mortality.
- Participant Treated With Rituximab and Radiation Only: Participant treated with rituximab and radiation only. Did not receive either interferon or etoposide/prednisone/vincristine/cyclophosphamide/doxorubicin/rituximab therapy.
- Participants Treated With Cross-over Interferon: Participants initially treated with etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (EPOCH-R) who relapse, or progress may crossover to receive interferon.
- Participants Treated With Cross-over EPOCH-R: Participants initially treated with Interferon who progress may crossover to receive etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin and rituximab (EPOCH-R).
Arm/Group | Participants Treated With Initial Interferon Therapy | Treated With Initial Etoposide,Prednisone,Vincristine,Cyclophosphamide,Doxorubicin,Rituximab Therapy | Participants Enrolled But Not Treated | Participant Treated With Rituximab and Radiation Only | Participants Treated With Cross-over Interferon | Participants Treated With Cross-over EPOCH-R
Number analyzed (Participants) | 60 | 28 | 5 | 1 | 10 | 24
Participants | 57 | 28 | 0 | 1 | 10 | 24

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored/assessed, up to a maximum of 27 years. Adverse Events were monitored/assessed from the first study intervention, Study Day 1 of Cycle 1 through 30 days after the study agent (s) was/were administered, up to a maximum of 49 months.
Description: All the deaths may not be accounted for in the serious and/or other adverse event tables since these were only collected during therapy and for 30 days following completion of therapy (as pre-specified in the protocol) whereas mortality data was collected up to a maximum of 27 years.
Arm/Group | Participants Treated With Initial Interferon Therapy | Treated With Initial Etoposide,Prednisone,Vincristine,Cyclophosphamide,Doxorubicin,Rituximab Therapy | Participants Enrolled But Not Treated | Participant Treated With Rituximab and Radiation Only | Participants Treated With Cross-over EPOCH-R | Participants Treated With Cross-over Interferon
All-Cause Mortality (participants affected / at risk) | 29/60 | 15/28 | 1/5 | 0/1 | 14/24 | 6/10
Serious Adverse Events (participants affected / at risk) | 21/60 | 20/28 | 0/5 | 0/1 | 15/24 | 6/10
Other Adverse Events (participants affected / at risk) | 57/60 | 28/28 | 0/5 | 1/1 | 24/24 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Treated With Initial Interferon Therapy (N=60) | Treated With Initial Etoposide,Prednisone,Vincristine,Cyclophosphamide,Doxorubicin,Rituximab Therapy (N=28) | Participants Enrolled But Not Treated (N=5) | Participant Treated With Rituximab and Radiation Only (N=1) | Participants Treated With Cross-over EPOCH-R (N=24) | Participants Treated With Cross-over Interferon (N=10)
ALT, SGPT (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Arrhythmia - Other (Specify, __): sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coagulation - Other (Specify, __): HPS (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death not associated with CTCAE term::Death NOS (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death not associated with CTCAE term::Disease progression NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Infections and infestations) | 10 (18) | 14 (34) | 0 (0) | 0 (0) | 10 (18) | 4 (8) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal - Other (Specify, __): Worsening GERD (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Bronchus
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Lung (pneumonia)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Urinary tract NOS
Infection - Other (Specify, __): Thyroid (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bladder (urinary) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bronchus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC::Lung (pneumonia) (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with unknown ANC::Rectum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Chest wall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis/thrombus/embolism (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Thrombotic microangiopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — (e.g., thrombotic thrombocytopenic purpura [TTP] or hemolytic uremic syndrome [HUS])
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Treated With Initial Interferon Therapy (N=60) | Treated With Initial Etoposide,Prednisone,Vincristine,Cyclophosphamide,Doxorubicin,Rituximab Therapy (N=28) | Participants Enrolled But Not Treated (N=5) | Participant Treated With Rituximab and Radiation Only (N=1) | Participants Treated With Cross-over EPOCH-R (N=24) | Participants Treated With Cross-over Interferon (N=10)
ALT, SGPT (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 35 (64) | 16 (32) | 0 (0) | 1 (1) | 17 (44) | 9 (23)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 34 (55) | 11 (21) | 0 (0) | 0 (0) | 18 (36) | 7 (15)
Albumin, serum-low (hypoalbuminemia) (Hepatobiliary disorders) | 32 (46) | 16 (31) | 0 (0) | 1 (1) | 17 (31) | 6 (12)
Alkaline phosphatase (Hepatobiliary disorders) | 27 (40) | 9 (11) | 0 (0) | 0 (0) | 15 (28) | 5 (6)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 6 (6) | 13 (16) | 0 (0) | 0 (0) | 3 (3) | 4 (6)
Allergy/Immunology - Other (Specify, __): perioral/ nasal fullness (Immune system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Anorexia (Gastrointestinal disorders) | 24 (30) | 14 (19) | 0 (0) | 0 (0) | 17 (22) | 7 (12)
Ataxia (incoordination) (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Auditory/Ear - Other (Specify, __): Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bilirubin (hyperbilirubinemia) (Hepatobiliary disorders) | 8 (14) | 6 (11) | 0 (0) | 0 (0) | 5 (10) | 3 (7)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 6 (6) | 4 (4) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 19 (31) | 10 (14) | 0 (0) | 0 (0) | 11 (21) | 5 (8)
Cheilitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coagulation - Other (Specify, __): HPS (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conduction abnormality/atrioventricular heart block::AV Block-Second degree Mobitz Type II (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 2 (5) | 2 (2) | 0 (0) | 0 (0) | 1 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 15 (19) | 16 (24) | 0 (0) | 0 (0) | 9 (11) | 7 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (22) | 11 (14) | 0 (0) | 0 (0) | 11 (12) | 6 (8)
Creatinine (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cushingoid appearance (e.g., moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 16 (30) | 14 (22) | 0 (0) | 0 (0) | 12 (26) | 6 (10)
Distension/bloating, abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 12 (13) | 12 (14) | 0 (0) | 0 (0) | 6 (7) | 6 (7)
Dry eye syndrome (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (5) | 4 (4) | 0 (0) | 0 (0) | 2 (3) | 3 (3)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 15 (18) | 14 (24) | 0 (0) | 0 (0) | 8 (11) | 8 (16)
Edema: limb (Blood and lymphatic system disorders) | 8 (13) | 9 (12) | 0 (0) | 0 (0) | 5 (10) | 4 (6)
Erectile dysfunction (Reproductive system and breast disorders) | 7 (7) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 48 (75) | 25 (62) | 0 (0) | 0 (0) | 22 (44) | 10 (32)
Febrile neutropenia (Infections and infestations) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 34 (45) | 15 (28) | 0 (0) | 0 (0) | 16 (27) | 7 (17)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
GGT (gamma-Glutamyl transpeptidase) (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 20 (40) | 18 (41) | 0 (0) | 1 (1) | 12 (30) | 6 (16)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 14 (21) | 15 (18) | 0 (0) | 0 (0) | 13 (20) | 6 (7)
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 6 (6) | 5 (5) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Hemoglobin (Renal and urinary disorders) | 38 (92) | 25 (86) | 0 (0) | 1 (1) | 18 (70) | 9 (29)
Hemorrhage, CNS (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hemorrhage, GU::Urinary NOS (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hemorrhage, pulmonary/upper respiratory::Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (5) | 0 (0) | 0 (0) | 2 (2) | 2 (4)
Hemorrhage, pulmonary/upper respiratory::Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flashes/flushes (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 6 (7) | 3 (7) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Ileus, GI (functional obstruction of bowel, i.e., neuro-constipation) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incontinence, anal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Blood
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Bronchus
Infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Colon
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Lip/perioral
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Lung (pneumonia)
Infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Mucosa
Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Oral cavity-gums (gingivitis)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Skin (cellulites)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Upper aerodigestive NOS
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Urethra
Infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) — (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)::Urinary tract NOS
Infection - Other (Specify, __): Fingernail (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Specify, __): Giardia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Specify, __): Shingles (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection - Other (Specify, __): ingrown nail (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection - Other (Specify, __): r/t PICC (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (Specify, __): thrush, URI, inner ear (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bladder (urinary) (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Blood (Infections and infestations) | 3 (3) | 2 (4) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bronchus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Colon (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Dental-tooth (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::External ear (otitis externa) (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Eye NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lip/perioral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 4 (6) | 3 (3) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Mucosa (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Neck NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Nerve-peripheral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Peritoneal cavity (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Rectum (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper aerodigestive NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 7 (8) | 1 (1) | 0 (0) | 0 (0) | 5 (6) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Infections and infestations) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Vagina (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Vein (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC::Anal/perianal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with unknown ANC::Bronchus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with unknown ANC::Mucosa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Insomnia (Nervous system disorders) | 18 (22) | 7 (7) | 0 (0) | 0 (0) | 10 (14) | 2 (2)
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 40 (131) | 25 (106) | 0 (0) | 1 (1) | 19 (105) | 8 (36)
Leukoencephalopathy (radiographic findings) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 38 (70) | 21 (64) | 0 (0) | 1 (1) | 17 (49) | 8 (20)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 13 (26) | 7 (11) | 0 (0) | 0 (0) | 9 (22) | 4 (7)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 11 (17) | 11 (22) | 0 (0) | 0 (0) | 7 (13) | 3 (5)
Memory impairment (Nervous system disorders) | 7 (7) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Mood alteration::Agitation (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mood alteration::Anxiety (Nervous system disorders) | 6 (7) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Mood alteration::Depression (Nervous system disorders) | 20 (22) | 6 (8) | 0 (0) | 0 (0) | 8 (8) | 5 (7)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 16 (40) | 19 (42) | 0 (0) | 0 (0) | 16 (40) | 8 (24)
Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 1 (1) | 2 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis/stomatitis (functional/symptomatic)::Pharynx (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy)::Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy)::Whole body/generalized (Musculoskeletal and connective tissue disorders) | 5 (7) | 12 (12) | 0 (0) | 0 (0) | 4 (6) | 5 (5)
Musculoskeletal/Soft Tissue - Other (Specify, __): Fracture-L humerus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 26 (33) | 17 (29) | 0 (0) | 0 (0) | 12 (16) | 8 (15)
Neurology - Other (Specify, __): Increased peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurology - Other (Specify, __): Increased peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurology - Other (Specify, __): Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0
Neuropathy: cranial::CN II Vision (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 9 (10) | 3 (4) | 0 (0) | 0 (0) | 7 (8) | 1 (2)
Neuropathy: sensory (Nervous system disorders) | 22 (30) | 19 (33) | 0 (0) | 0 (0) | 14 (22) | 8 (18)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 36 (119) | 25 (91) | 0 (0) | 1 (1) | 20 (102) | 8 (32)
Ocular/Visual - Other (Specify, __): b/l optic neuritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis, middle ear (non-infectious) (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 6 (6) | 3 (5) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Pain - Other (Specify, __): Injection Site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain - Other (Specify, __): Injection site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain - Other (Specify, __): PICC site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain::Abdomen NOS (Gastrointestinal disorders) | 9 (10) | 2 (3) | 0 (0) | 0 (0) | 5 (6) | 2 (3)
Pain::Anus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain::Back (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 9 (16) | 14 (27) | 0 (0) | 0 (0) | 8 (15) | 5 (10)
Pain::Cardiac/heart (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Chest wall (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain::Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Pain::Dental/teeth/periodontal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::External ear (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain::Extremity-limb (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain::Face (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Head/headache (Nervous system disorders) | 22 (28) | 13 (19) | 0 (0) | 0 (0) | 8 (13) | 7 (11)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 13 (16) | 2 (6) | 0 (0) | 0 (0) | 8 (10) | 2 (6)
Pain::Kidney (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain::Middle ear (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 23 (32) | 8 (14) | 0 (0) | 0 (0) | 11 (16) | 5 (11)
Pain::Neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Neuralgia/peripheral nerve (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain::Pelvis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain::Testicle (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Throat/pharynx/larynx (Gastrointestinal disorders) | 3 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain::Urethra (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Personality/behavioral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 6 (8) | 5 (7) | 0 (0) | 0 (0) | 2 (4) | 2 (2)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 38 (95) | 26 (106) | 0 (0) | 1 (1) | 20 (76) | 9 (38)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 5 (5) | 3 (5) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 12 (17) | 6 (14) | 0 (0) | 0 (0) | 7 (12) | 4 (8)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pulmonary/Upper Respiratory - Other (Specify, __): INFECTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify, __): Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 10 (13) | 8 (13) | 0 (0) | 0 (0) | 7 (8) | 5 (8)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash: dermatitis associated with radiation::Radiation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal/Genitourinary - Other (Specify, __): Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rigors/chills (General disorders) | 22 (26) | 10 (12) | 0 (0) | 0 (0) | 11 (14) | 8 (10)
Secondary Malignancy - possibly related to cancer treatment (Specify, __) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 13 (19) | 3 (3) | 0 (0) | 0 (0) | 7 (12) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 15 (20) | 16 (33) | 0 (0) | 0 (0) | 11 (15) | 6 (19)
Somnolence/depressed level of consciousness (Nervous system disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Supraventricular and nodal arrhythmia::Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 5 (5) | 4 (4) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Supraventricular and nodal arrhythmia::Supraventricular arrhythmia NOS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sweating (diaphoresis) (General disorders) | 8 (9) | 7 (7) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Syncope (fainting) (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 11 (13) | 9 (11) | 0 (0) | 0 (0) | 8 (10) | 5 (6)
Thrombosis/embolism (vascular access-related) (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis/thrombus/embolism (Cardiac disorders) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular - Other (Specify, __): Thromboembolic event (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia::Ventricular arrhythmia NOS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision-blurred vision (Eye disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision-photophobia (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 13 (22) | 13 (20) | 0 (0) | 0 (0) | 8 (14) | 6 (11)
Watery eye (epiphora, tearing) (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight gain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight loss (General disorders) | 19 (21) | 5 (6) | 0 (0) | 0 (0) | 11 (13) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT00001379/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT00001379/ICF_001.pdf